CLINICAL TRIAL: NCT03589703
Title: Management of Chronic Low Back Pain in Older Adults Using Auricular Point Acupressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Constance Johnson, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-SN-21-1059; 1R01AG056587-01A1 (NIH)
Record Dates: First submitted 2018-05-22; First posted 2018-07-18 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic Low Back Pain; cLBP; pain; acupressure
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T-APA (Active Comparator): Patients with active points related to cLBP. Will receive acupressure within the two zones for cLBP located on the front and back of the ear and three points known for alleviating stress and pain.
  Interventions: Other: Target ear points related to chronic low back pain (T-APA)
- NT-APA (Active Comparator): The same procedure for APA will be applied but the tapes/seeds will be placed on five different ear points, comprising mouth, stomach, duodenum, internal ear, and tonsil.
  These points are chosen for the non-target ear points of APA treatment for two reasons. First, they are distinct from the zones of the ear (and the points therein) associated with the lower back, and correspond to body regions in which the participant is usually pain-free. Second, they are equivalent in number to those points used in the APA treatment group.
  Interventions: Other: Non-Target ear Points not related to chronic low back pain (NT-APA)
- Enhanced Educational Control Group (CG-2) (Other): Participants in the enhanced educational control group will be given the cLBP educational booklet and visit the office weekly for assessment (i.e., blood draws and questionnaires), which is the same schedule as that for the APA groups.
  Interventions: Other: Enhanced Educational Control Group (CG-2)

INTERVENTIONS:
Other: Target ear points related to chronic low back pain (T-APA) — Light touch using vaccaria seeds on specific points of the ear.
  Arms: T-APA
Other: Non-Target ear Points not related to chronic low back pain (NT-APA) — Light touch using vaccaria seeds on different points of the ear (compared to the APA group).
  Arms: NT-APA
Other: Enhanced Educational Control Group (CG-2) — No contact with the subject. Participants in the enhanced educational control group will be given the cLBP educational booklet.
  Arms: Enhanced Educational Control Group (CG-2)

SUMMARY:
Almost one-third (30%) of persons 60 years and older suffer from cLBP and cause a significant negative impact on individuals and society in the U.S. The goal of managing cLBP is decreased pain and disability.To accomplish this, cLBP sufferers often use analgesics including opioids to decrease pain and facilitate activity, but the side effects caused by these medications are problematic. A better pain management strategy clearly needs to be developed.

The investigators propose to test auricular point acupressure (APA), a non-invasive, easily administered, patient-controlled, and non-pharmacological strategy, to provide rapid, safe, and an innovative solution for chronic low back pain (cLBP) in older adults. APA involves an acupuncture-like stimulation of the ear without needles. With APA, small seeds are taped to specific ear points. The patient is taught to apply pressure to the seeds, with the thumb and index finger, three times a day (morning, noon, and evening) for three minutes each session to achieve pain relief. The investigators have developed a detailed APA protocol to teach health-care providers without experience in acupuncture and traditional Chinese Medicine that investigators can learn about APA in brief educational seminars as a treatment including the systematic identification of ear points (called auricular diagnosis). The investigators teach methods that enable patients to continue using APA to self-manage participants' pain.

Brain imaging studies in acupuncture indicate that acupuncture can restore normal functional connectivity related to pain reduction. Studies suggest that stimulation of ear points (1) excites the somatotopic reflex system in the brain and that pathological brain patterns are electrically reset to stop the unwanted activation of spinal pain pathways, explaining the possible immediate pain relief that patients feel after APA and (2) cause a broad spectrum of systemic effects, such as vasodilation, by releasing endorphin to elicit short-term analgesic effects or neuropeptide-induced anti-inflammatory cytokines, which may explain long-term effects.

The Ecological Momentary Assessment (EMA) smart phone app will be used to collect real-time cLBP outcomes and adherence to APA practice. Treatment and nonspecific psychological placebo effects will be measured via questionnaires for all participants. Neuro-transmitters is measured by inflammatory biomarkers. Blood samples will be collected for serum collection and a multiplex bead-based immunofluorescence assay performed to check for serum levels. Mini-Mental State Examination will be used to screen for cognitive function, also HRQoL, satisfaction, treatment beliefs and expectations, sleep, relaxation effects, catastrophizing and fear/avoidance, and placebo effects will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* Able to read and write English
* cLBP that has persisted at least 3 months and has pain on at least half of the days for the previous 6 months
* Average intensity of pain ≥ 4 on a 11-point numerical pain scale in the previous week
* Have intact cognition (Mini-Mental State Examination (MMSE) > 24)
* Willing to commit to up to 13-17 months as a study participant, depending on which group the participant is placed in
* Able to apply pressure to the seeds with tapes on their ears

Exclusion Criteria:

* Malignant or autoimmune diseases (e.g., rheumatoid arthritis), in which the pain from the disease cannot be separated from the low back pain by the participant
* Known acute compression fractures caused by osteoporosis, spinal stenosis, spondylolysis, or spondylolisthesis because these conditions may confound treatment effects or the interpretation of results
* Sciatica with leg pain greater than back pain
* Allergy to the tape
* Use of some types of hearing aids (size may obstruct the placement of seeds)
* Pain in other parts of the body that is more severe than the cLBP and which occurs daily or almost every day with at least moderate intensity or acute pain
* Neurological disorders that could interfere with pain reporting or confound performance on the other outcomes, cerebral tumor, Alzheimer's disease (or other cognitive illnesses), prior stroke, or multiple sclerosis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2023-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constance Johnson, PhD, MS, RN, Principal Investigator — The University of Texas Health Science Center, Houston; Nada Lukkahatai, PhD, MSN, RN, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - The University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang J, Castelli G, Shen A, Li J, Kawi J, Wu H, Christo P, Campbell CM, Thrul J, Johnson CM, Lukkahatai N. Effectiveness of acupressure at different ear acupoints on Insomnia: A secondary analysis of a randomized controlled trial. Sleep Med X. 2025 Oct 15;10:100158. doi: 10.1016/j.sleepx.2025.100158. eCollection 2025 Dec 15. PMID 41170529
- [Derived] Kawi J, Yeh CH, Lukkahatai N, Wu H, Morone NE, Glick R, Schlenk EA, Campbell C, Thrul J, Huang X, Wang H, Jia HM, Christo P, Johnson C. Auricular point acupressure for older adults with chronic low back pain: a randomized controlled trial. Pain Med. 2025 Sep 1;26(9):515-526. doi: 10.1093/pm/pnaf035. PMID 40152243
- [Derived] Yeh CH, Li C, Glick R, Schlenk EA, Albers K, Suen LK, Lukkahatai N, Salen N, Pandiri S, Ma W, Perrin N, Morone NE, Christo PJ. A prospective randomized controlled study of auricular point acupressure to manage chronic low back pain in older adults: study protocol. Trials. 2020 Jan 20;21(1):99. doi: 10.1186/s13063-019-4016-x. PMID 31959226

RESULTS

PARTICIPANT FLOW:
Groups:
- T-APA: Patients with active points related to chronic lower back pain (cLBP) will receive acupressure within the two zones for cLBP located on the front and back of the ear and three points known for alleviating stress and pain.
  Target ear points related to chronic low back pain (T-APA): Light touch using vaccaria seeds on specific points of the ear.
- NT-APA: The same procedure for APA will be applied but the tapes/seeds will be placed on five different ear points, comprising mouth, stomach, duodenum, internal ear, and tonsil.
  These points are chosen for the non-target ear points of APA treatment for two reasons. First, they are distinct from the zones of the ear (and the points therein) associated with the lower back, and correspond to body regions in which the participant is usually pain-free. Second, they are equivalent in number to those points used in the APA treatment group.
  Non-Target ear Points not related to chronic low back pain (NT-APA): Light touch using vaccaria seeds on different points of the ear (compared to the APA group).
Period: Overall Study
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Started | 92 | 91 | 89
Completed Follow up 1 Month Post-intervention | 81 | 68 | 71
Completed | 81 | 68 | 71
Not Completed | 11 | 23 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2) | Total
Number analyzed (Participants) | 92 | 91 | 89 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (6.5) | 68.7 (7.1) | 71.1 (7.2) | 70.0 (7.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 59 | 56 | 59 | 174
  Male | 32 | 35 | 29 | 96
  Unknown or Not Reported | 1 | 0 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 84 | 67 | 67 | 218
  Unknown or Not Reported | 7 | 23 | 20 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 51 | 58 | 55 | 164
  White | 39 | 28 | 30 | 97
  More than one race | 1 | 2 | 0 | 3
  Unknown or Not Reported | 1 | 1 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 92 | 91 | 89 | 272
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) is calculated as weight in kilograms divided by the square of height in meters.
  kg/m^2 | 31.3 (8.5) | 31.1 (7.7) | 30.6 (7.0) | 31.0 (7.7)
Education Level [Count of Participants; unit: Participants]
  High School or Less | 27 | 36 | 37 | 100
  Some College | 20 | 17 | 11 | 48
  College or Higher | 45 | 38 | 41 | 124
Employment Status [Count of Participants; unit: Participants]
  Employed | 9 | 11 | 13 | 33
  Unemployed or Retired | 80 | 79 | 75 | 234
  Unknown | 3 | 1 | 1 | 5
Severity of Comorbidity as Assessed by Charlson Comorbidity Index [Mean (Standard Deviation); unit: score on a scale] — Total score on the Charlson Comorbidity Index is 0 to 37. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use.
  score on a scale | 1.3 (2.8) | 1.0 (2.2) | 1.0 (1.6) | 1.1 (2.2)
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 15 | 21 | 11 | 47
  Never Smoked | 38 | 26 | 39 | 103
  Previously Smoked | 39 | 44 | 39 | 122

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity as Assessed by the Numeric Rating Scale (NRS)
Description: Pain intensity as assessed by the NRS for worst pain in the past 7 days using a 0-10 scale (0 = "no pain" and 10 = "worst pain imaginable")
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 92 | 91 | 89
score on a scale | 7.4 (1.7) | 7.0 (1.8) | 7.3 (1.7)

2. Primary Outcome: Pain Intensity as Assessed by the Numeric Rating Scale (NRS)
Description: as for outcome 1
Time Frame: 1 month post completion of the treatment (2 months after baseline)
Population: Data were not collected for 11 in the T-APA arm, 19 in the NT-APA arm, and 20 in the Control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 81 | 72 | 69
score on a scale | 5.6 (2.7) | 5.3 (2.7) | 6.6 (2.2)

3. Primary Outcome: Pain Interference as Assessed by the Brief Pain Inventory-short Form Pain Interference Subscale
Description: Pain interference is assessed by the Brief Pain Inventory pain interference subscale, which uses a 0-10 scale (0 = "does not interfere" and 10 = "completely interferes").
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 92 | 91 | 89
score on a scale | 3.2 (1.7) | 3.3 (1.7) | 3.1 (1.6)

4. Primary Outcome: Pain Interference as Assessed by the Brief Pain Inventory-short Form Pain Interference Subscale
Description: as for outcome 3
Time Frame: 1 month post completion of the treatment (2 months after baseline)
Population: Data were not collected for 11 in the T-APA arm, 19 in the NT-APA arm, and 20 in the Control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 81 | 72 | 69
score on a scale | 2.7 (1.9) | 2.5 (1.6) | 2.9 (1.7)

5. Primary Outcome: Physical Function as Assessed by the Roland Morris Disability Questionnaire (RMDQ)
Description: The Roland Morris Disability Questionnaire (RMDQ), 24-item measure, is used to assess the impact of back pain on their daily functioning. The score ranges from 0 (no disability) to 24 (maximum disability).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 92 | 91 | 89
score on a scale | 12.4 (5.3) | 12.6 (6.2) | 12.0 (5.9)

6. Primary Outcome: Physical Function as Assessed by the Roland Morris Disability Questionnaire (RMDQ)
Description: as for outcome 5
Time Frame: 1 month post completion of the treatment (2 months after baseline)
Population: Data were not collected for 11 in the T-APA arm, 19 in the NT-APA arm, and 18 in the Control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 81 | 72 | 71
score on a scale | 9.8 (6.2) | 9.6 (6.6) | 10.5 (5.8)

7. Secondary Outcome: Number of Participants Who Use Opioids
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 92 | 91 | 89
Participants | 44 | 45 | 32

8. Secondary Outcome: Number of Participants Who Use Opioids
Time Frame: 1 month post completion of the treatment (2 months after baseline)
Population: Data were not collected for 17 in the T-APA arm, 29 in the NT-APA arm, and 20 in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 75 | 62 | 69
Participants | 25 | 22 | 17

9. Secondary Outcome: APA Treatment Satisfaction as Assessed by Satisfaction Survey
Description: Satisfaction is assessed using a 5-point numeric rating scale:
  1. - Completely satisfied
  2. - Somewhat satisfied
  3. - Neither satisfied nor dissatisfied
  4. - Somewhat dissatisfied
  5. - Very dissatisfied
Time Frame: immediately post intervention (1 month after baseline)
Population: Data were not collected for 11 in the T-APA arm and 17 in the NT-APA arm. These data were not collected for any of the 89 in the control arm, as they did not receive the APA treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 81 | 74 | 0
score on a scale | 2.04 (0.993) | 2.16 (1.047) |

10. Secondary Outcome: APA Treatment Satisfaction as Assessed by Satisfaction Survey
Description: as for outcome 9
Time Frame: 1 month post completion of the treatment (2 months after baseline)
Population: Data were not collected for 17 in the T-APA arm and 29 in the NT-APA arm. These data were not collected for any of the 89 in the control arm, as they did not receive the APA treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 75 | 62 | 0
score on a scale | 2.29 (1.088) | 2.10 (0.953) |

11. Secondary Outcome: Quality of Life as Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS-29) - Anxiety
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS-29) is a 29-item profile instrument that can be used to assess seven subscales of health quality of life (QOL) for each of 7 domains-this outcome measure reports one of the 7 domains, anxiety. The raw score on the anxiety subscale is converted to a standardized T-score. T-score is reported here, and it ranges from 0 to 100, with a higher PROMIS T-score representing more of the concept being measured, that is, greater anxiety. PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population; therefore, an anxiety T-score of 40 is one SD better than average in terms of anxiety. A T-score below 55 is indicative of anxiety within normal limits.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 92 | 91 | 89
T-score | 51.0 (8.9) | 53.1 (10.8) | 51.8 (9.9)

12. Secondary Outcome: Quality of Life as Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS-29) - Anxiety
Description: as for outcome 11
Time Frame: 1 month post completion of the treatment (2 months after baseline)
Population: Data were not collected for 11 in the T-APA arm, 19 in the NT-APA arm, and 20 in the Control arm.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 81 | 72 | 69
T-score | 49.0 (9.5) | 48.8 (9.4) | 51.5 (10.0)

13. Secondary Outcome: Quality of Life as Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS-29) - Depression
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS-29) is a 29-item profile instrument that can be used to assess seven subscales of health quality of life (QOL) for each of 7 domains-this outcome measure reports one of the 7 domains, depression. The raw score on the depression subscale is converted to a standardized T-score. T-score is reported here, and it ranges from 0 to 100, with a higher PROMIS T-score representing more of the concept being measured, that is, greater depression. PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population; therefore, a depression T-score of 40 is one SD better than average in terms of depression. A T-score below 55 is indicative of depression within normal limits.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 92 | 91 | 89
T-score | 50.3 (9.6) | 52.7 (9.0) | 50.5 (9.1)

14. Secondary Outcome: Quality of Life as Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS-29) - Depression
Description: as for outcome 13
Time Frame: 1 month post completion of the treatment (2 months after baseline)
Population: Data were not collected for 11 in the T-APA arm, 19 in the NT-APA arm, and 20 in the Control arm.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 81 | 72 | 69
T-score | 49.1 (8.7) | 48.9 (8.3) | 49.6 (9.6)

15. Secondary Outcome: Quality of Life as Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS-29) - Sleep Disturbance
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS-29) is a 29-item profile instrument that can be used to assess seven subscales of health quality of life (QOL) for each of 7 domains-this outcome measure reports one of the 7 domains, sleep disturbance. The raw score on the sleep disturbance subscale is converted to a standardized T-score. T-score is reported here, and it ranges from 0 to 100, with a higher PROMIS T-score representing more of the concept being measured, that is, greater sleep disturbance. PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population; therefore, a sleep disturbance T-score of 40 is one SD better than average in terms of sleep disturbance. A T-score below 55 is indicative of sleep disturbance within normal limits.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 92 | 91 | 89
T-score | 56.0 (4.1) | 56.0 (3.3) | 55.5 (4.0)

16. Secondary Outcome: Quality of Life as Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS-29) - Sleep Disturbance
Description: as for outcome 15
Time Frame: 1 month post completion of the treatment (2 months after baseline)
Population: Data were not collected for 11 in the T-APA arm, 19 in the NT-APA arm, and 20 in the Control arm.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 81 | 72 | 69
T-score | 55.3 (3.4) | 55.9 (5.0) | 55.9 (3.3)

17. Secondary Outcome: Fear-Avoidance as Assessed by the Fear-avoidance Beliefs Questionnaire (FABQ)
Description: The fear-avoidance beliefs questionnaire (FABQ) focuses on participant's beliefs about how physical activity and work affect their pain. The questionnaire consists of 16 items in which a participant rates their agreement with each statement on a 7-point Likert scale where 0 = completely disagree and 6 =completely agree. The total score ranges from 0 to 96. A higher score indicates more strongly held fear-avoidance beliefs.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 92 | 91 | 89
score on a scale | 15.7 (8.3) | 17.0 (8.8) | 15.6 (8.6)

18. Secondary Outcome: Fear-Avoidance as Assessed by the Fear-avoidance Beliefs Questionnaire (FABQ)
Description: as for outcome 17
Time Frame: 1 month post completion of the treatment (2 months after baseline)
Population: Data were not collected for 11 in the T-APA arm, 29 in the NT-APA arm, and 21 in the Control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 81 | 62 | 68
score on a scale | 13.4 (9.0) | 14.8 (8.8) | 15.2 (8.4)

19. Secondary Outcome: Pain Catastrophizing as Assessed by the Pain Catastrophizing Scale (PCS)
Description: The PCS was included to detect exaggerated and negative interpretations of pain. It is a self-report scale that consists of13 items. Participants were asked to reflect on past painful experiences and to indicate to which degree he/she experienced symptoms such as helplessness or rumination when feeling pain. This is a 0-4 Likert scale (score sum 0-52) with responses ranging from "not at all" to "all the time," with higher scores indicate stronger catastrophizing.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 92 | 91 | 89
score on a scale | 15.7 (12.4) | 19.1 (14.2) | 15.9 (12.4)

20. Secondary Outcome: Pain Catastrophizing as Assessed by the Pain Catastrophizing Scale (PCS)
Description: as for outcome 19
Time Frame: 1 month post completion of the treatment (2 months after baseline)
Population: Data were not collected for 11 in the T-APA arm, 19 in the NT-APA arm, and 21 in the Control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 81 | 72 | 68
score on a scale | 14.1 (12.7) | 13.9 (11.8) | 13.8 (12.7)

21. Secondary Outcome: Memory as Assessed by the Stroop Test
Description: T-score will be reported, with a range of 0-100, with a higher score indicating better memory.
Time Frame: Baseline
Population: Data were not collected from any participant for this outcome measure.
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: Memory as Assessed by the Stroop Test
Description: T-score will be reported, with a range of 0-100, with a higher score indicating better memory.
Time Frame: 1 month post completion of the treatment (2 months after baseline)
Population: Data were not collected from any participant for this outcome measure.
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 0 | 0 | 0

23. Secondary Outcome: Relaxation as Assessed by Relaxation Response
Time Frame: Baseline
Population: Data were not collected from any participant for this outcome measure.
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 0 | 0 | 0

24. Secondary Outcome: Relaxation as Assessed by Relaxation Response
Time Frame: 1 month post completion of the treatment (2 months after baseline)
Population: Data were not collected from any participant for this outcome measure.
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: from start of intervention to end of intervention (4 weeks)
Arm/Group | T-APA | NT-APA | Enhanced Educational Control Group (CG-2)
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/91 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/91 | 0/89
Other Adverse Events (participants affected / at risk) | 69/92 | 48/91 | 0/89
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-APA (N=92) | NT-APA (N=91) | Enhanced Educational Control Group (CG-2) (N=89)
Itching/Discomfort on the ear where the seed was placed (General disorders) | 69 (183) | 48 (112) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT03589703/Prot_SAP_000.pdf